CLINICAL TRIAL: NCT01898312
Title: The Effect of a Progesterone Receptor Modulator on Breast Tissue in Women With BRCA-1 and -2 Mutations - a Placebo Controlled RCT.
Brief Title: BRCA1/2 and Effect of Mifepristone on the Breast
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, MD Ph.D, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2012-003703-35
Record Dates: First submitted 2013-07-05; First posted 2013-07-12 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Women With Mutations in the Breast Cancer Susceptibility Genes BRCA1,2
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mifepristone (Experimental): treatment with oral mifepristone 50 mg every second day for 12 weeks in 30 women with BRCA 1 or 2 mutation
  Interventions: Drug: Mifepristone
- TrioBe (Placebo Comparator): treatment with a quarter of a tablet of TrioBe every second day for 12 weeks
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Randomised controlled trial of Mifepristone and placebo comparator Triobe

SUMMARY:
Ovarian steroids, as well as their synthetic counterparts gestagens and estrogens have a role in breast cell proliferation and the development of breast cancer. Here, the effect of a progesterone receptor modulator, mifepristone, on cell proliferation in human breast tissue in vivo will be studied in women with BRCA-1 or -2 mutations. Our preliminary results implicate a possible protective effect of mifepristone in breast epithelium. The ability of mifepristone to block breast epithelial cell proliferation may prevent tumorigenesis and may also prove beneficial when used for contraceptive purposes and on other indications. The proposed project concerns a Randomized Controlled Trial on mifepristone versus placebo treatment of women with BRCA-1or -2 mutations with a high risk/incidence of breast cancer and ovarian cancer.

DETAILED DESCRIPTION:
Objectives • Research objective To study the safety and effect of treatment with mifepristone, a progesterone receptor modulator, on epithelial cell proliferation in human breast tissue in women with BRCA-1 or -2 mutations prior to protective mastectomy.

Project description

• Hypothesis/ Theory Mifepristone treatment exerts an antiproliferative, protective effect on breast tissue in women with BRCA-1 or -2 mutations

Study Design Randomized, double blind, placebo controlled trial. Women will be recruited among patients with BRCA-1 or -2 mutations scheduled for prophylactic mastectomy. Included women will be randomized to a 3-month treatment with mifepristone, 50 mg (Mifegyne, Exelgyn, Paris, France) or placebo taken orally every second day. Breast biopsies will be obtained in the luteal phase prior to start of treatment and again during surgery.

ELIGIBILITY:
Inclusion criteria:

* Pre-menopausal women, >/= 18 years of age
* with good general health and
* regular menstrual cycles (25-35 days) who are willing and
* able to participate after giving informed consent.
* women having BRCA1/2 mutation and have decided to undergo risk reducing mastectomy

Exclusion criteria includes:

* Any hormonal treatment used within 2 months prior to study start and
* Any contraindication to mifepristone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
epithelial cell proliferation in breast tissue | 3 months
  Changes from baseline after 12 weeks of mifepristone treatment in epithelial cell proliferation by measuring expression of genes specifically in the pathways involving apoptotic and cell proliferation by microarray study, including PTEN, Bcl-2 and Ki-67 along with steroid receptors.

SECONDARY OUTCOMES:
Vital signs and safety lab analysis | 3 months
  Safety data includes vital signs, general- and gynecological-, incl breast - examinations, safety lab (hematology (blood status+CRP), kidney function (Na, K, krea) liver function (ASAT, ALAT, ALP, GT, bilirubin) , thyroid function (TSH,T3,T4), hormonal values FSH ,LH , PRL, SHBG, testosterone, E2 (sensitive) progesterone, urine dipstick and pregnancy test (prior to start). Endometrial histology will be investigated in biopsies obtained at baseline and at surgery. Women with BRCA-1/-2 mutations are followed according to the existing clinical routine with regard to ovarian cancer screening.
Side effects and Adverse Events | 3 months
  Side effects of mifepristone are mild and the only significant side effect reported in previous clinical trials with the same regimen has been mild flushes. All side effects and SAE/AE as well as any concomitant medication will be recoded by the participating patients in a dairy.
Endometrial effects | 3 months
  Bleeding patterns and endometrial morphologywill be studied. Endometrial histology and progesterone receptor modulator associated changes will be investigated in biopsies obtained at baseline and at surgery. Bleeding pattern will be registered during the study period by the participating women.
Ovarian effects | 3 months
  Women with BRCA-1/-2 mutations are followed according to the existing clinical routine with regard to ovarian cancer screening.
Breast symptom evaluation | 3months
  Breast symptom evaluation will be registered at baseline and during the study by a breast symptom score.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell Danielsson, Professor, Principal Investigator — Dept of Womens and Childrens Health Karolinska Institutet; Angelique Flöter Rådestad, MD PhD, Study Chair — Dept of Womens and Childrens Health, Karolinska Institutet
Locations (1):
- Department of Woman and Child Health Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Engman M, Skoog L, Soderqvist G, Gemzell-Danielsson K. The effect of mifepristone on breast cell proliferation in premenopausal women evaluated through fine needle aspiration cytology. Hum Reprod. 2008 Sep;23(9):2072-9. doi: 10.1093/humrep/den228. Epub 2008 Jun 24. PMID 18579510
- [Background] Isern AE, Loman N, Malina J, Olsson H, Ringberg A. Histopathological findings and follow-up after prophylactic mastectomy and immediate breast reconstruction in 100 women from families with hereditary breast cancer. Eur J Surg Oncol. 2008 Oct;34(10):1148-54. doi: 10.1016/j.ejso.2008.03.002. Epub 2008 Apr 23. PMID 18434071
- [Background] Kauff ND, Brogi E, Scheuer L, Pathak DR, Borgen PI, Hudis CA, Offit K, Robson ME. Epithelial lesions in prophylactic mastectomy specimens from women with BRCA mutations. Cancer. 2003 Apr 1;97(7):1601-8. doi: 10.1002/cncr.11225. PMID 12655515
- [Background] Poole AJ, Li Y, Kim Y, Lin SC, Lee WH, Lee EY. Prevention of Brca1-mediated mammary tumorigenesis in mice by a progesterone antagonist. Science. 2006 Dec 1;314(5804):1467-70. doi: 10.1126/science.1130471. PMID 17138902
- [Derived] Bartlett TE, Evans I, Jones A, Barrett JE, Haran S, Reisel D, Papaikonomou K, Jones L, Herzog C, Pashayan N, Simoes BM, Clarke RB, Evans DG, Ghezelayagh TS, Ponandai-Srinivasan S, Boggavarapu NR, Lalitkumar PG, Howell SJ, Risques RA, Radestad AF, Dubeau L, Gemzell-Danielsson K, Widschwendter M. Antiprogestins reduce epigenetic field cancerization in breast tissue of young healthy women. Genome Med. 2022 Jun 15;14(1):64. doi: 10.1186/s13073-022-01063-5. PMID 35701800